CLINICAL TRIAL: NCT02583191
Title: CONKO_011/ AIO-SUP-0115/Ass.: Rivaroxaban in the Treatment of Venous Thromboembolism (VTE) in Cancer Patients - a Randomized Phase III Study
Brief Title: Rivaroxaban in the Treatment of Venous Thromboembolism (VTE) in Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment was not as expected.
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Charite University, Berlin, Germany (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONKO-011 AIO-SUP-0115/ass.
Record Dates: First submitted 2015-10-15; First posted 2015-10-22 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Venous Thromboembolism; Cancer
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental): Arm A: Rivaroxaban
  Interventions: Drug: Rivaroxaban
- low-molecular heparine (Active Comparator): Arm B: standard treatment with low-molecular heparine
  Interventions: Drug: low-molecular heparine

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban 15 mg twice daily for 21 days, followed by 20 mg once daily over a period of 3 months
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: low-molecular heparine — LMWH in therapeutic dosage (1-2× daily s.c.) according to standards of the individual study center, using licensed dosages, e.g.
  * Enoxaparin 1 mg/kg BW twice daily
  * Tinzaparin 175 I.E./kg BW once daily
  * Dalteparin 200 I.E./kg BW once daily
  Arms: low-molecular heparine

SUMMARY:
The purpose of this study is to show feasibility (efficacy and safety) of Rivaroxaban in the treatment of VTE in cancer patients in comparison to the standard treatment with low molecular weight heparin (LMWH).

Tumor patients with active cancer and newly diagnosed thromboembolic events are randomised to receive either Rivaroxaban or the standard treatment with low-molecular heparin.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and objectively confirmed acute venous thromboembolism
* Active malignancy
* Life expectancy of at least 6 months
* Performance-Status according to Karnofsky Performance Scale ≥ 70 %
* Patient's compliance and geographical situation allowing an adequate follow up
* platelets ≥ 100.000 /μl, INR < 1.5, PTT < 40 sec.
* written informed consent of the patient prior to any procedure in connection with the study
* male and female patients with an age of at least 18 years

Exclusion Criteria:

* therapeutic anticoagulation > 96 hours prior to study treatment
* known allergic reactions against the study drugs or the substances included therein
* known conditions associated with high risk of bleeding, known history of hemorrhagic diathesis
* acute clinically relevant bleeding in the last 2 weeks
* any history of spontaneous major/cerebral bleeding
* history of heparin induced thrombocytopenia II
* pregnant or breast-feeding women. Women of child-bearing potential must have a negative pregnancy test performed < 7 days prior to start of the treatment
* severe renal insufficiency (GFR < 30 ml/min)
* liver disease with coagulation impairment, including Child B and C
* cirrhosis
* acute medical illness
* treatment of the underlying cancer with experimental therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Patient-reported treatment satisfaction (convenience) with Rivaroxaban in the treatment of acute VTE in cancer patients in comparison with the standard treatment with low molecular weight heparin | From randomization to 4 weeks after treatment start

SECONDARY OUTCOMES:
Rate of symptomatic venous thrombembolism-recurrence within 3 months exploratory analysis for patients with treatment | From randomization to 3 months after treatment start
Exploratory analysis for "time on treatment" | From randomization to 12 weeks after treatment start
Subgroup analysis with regard to rate of Pulmonary embolism, venous thrombembolism recurrence and bleedings (major, clinically relevant, minor) according to stratification characteristics | From randomization to end of follow up (up to 24 weeks)
Rate of myocardial infarction and ischemic stroke | From randomization to end of follow up (up to 24 weeks)
Compliance of patients (adherence) | From randomization to end of follow up (up to 24 weeks)
Overall mortality 3 and 6 months after randomization | From randomization to 3 and 6 months after randomization
Quality of Life (Spitzer Index (Spitzer 1981), Anticlot Treatment Scale (ACTS) and TSQM | 4 weekly, up to 12 weeks
Rate of clinically relevant bleeding (major + clinically relevant non major) within 3 months | From randomization to 3 months after randomization
Rate of minor bleedings within 3 months | From randomization to 3 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinik, Aachen, Germany

REFERENCES:
- [Derived] Riaz IB, Fuentes HE, Naqvi SAA, He H, Sipra QR, Tafur AJ, Padranos L, Wysokinski WE, Marshall AL, Vandvik PO, Montori V, Bryce AH, Liu H, Badgett RG, Murad MH, McBane RD 2nd. Direct Oral Anticoagulants Compared With Dalteparin for Treatment of Cancer-Associated Thrombosis: A Living, Interactive Systematic Review and Network Meta-analysis. Mayo Clin Proc. 2022 Feb;97(2):308-324. doi: 10.1016/j.mayocp.2020.10.041. Epub 2021 Jun 22. PMID 34172290